CLINICAL TRIAL: NCT03069339
Title: Carvedilol, Endoscopic Variceal Ligation or Combination of Both for Prevention of First Variceal Bleed in Child's B & C Cirrhosis: A Randomized Controlled Trial
Brief Title: Carvedilol, Endoscopic Variceal Ligation or Combination of Both for Prevention of First Variceal Bleed in Child's B & C Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-07
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carvedilol+EVL (Experimental)
  Interventions: Drug: Carvedilol; Procedure: Endoscopic Variceal Ligation
- Carvedilol (Experimental)
  Interventions: Drug: Carvedilol
- EVL (Active Comparator)
  Interventions: Procedure: Endoscopic Variceal Ligation

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will start at starting dose of 3.125 mg BD followed by 6.25 mg BD followed by 12.5 mg BD if BP 90/60 mmHg and HR 55/min
  Arms: Carvedilol; Carvedilol+EVL
Procedure: Endoscopic Variceal Ligation — EVL will be done every 3 weeks till eradication
  Arms: Carvedilol+EVL; EVL

SUMMARY:
Study Design: Open labeled randomized controlled trial. The study will be conducted on patients attending outpatient or admitted to admitted to Department of Hepatology from January 2017 to December 2018 at ILBS, New Delhi

ELIGIBILITY:
Inclusion Criteria:

* Liver Cirrhotics between 18-70 yrs of age (cirrhosis diagnosed on the basis of clinical, biochemical, fibroscan & imaging.)
* CTP ≥ 7-15 (Child's B/C)
* Small esophageal varices with RCS and large esophageal varices (>5 mm)
* No history of previous bleed

Exclusion Criteria:

* Malignancy-HCC, PVT
* Child A
* MELD >35
* Contraindications to β blockers.
* Platelet count < 30,000/mm3
* Previous endoscopic variceal treatment. (Beyond 21 days)
* Patients having an indication for TIPS or requiring more than 1 therapeutic ascitic tapping/month
* Post TIPS, Shunt surgery
* Acute kidney injury (Sr.Cr>1.5mg/dl)
* Non cirrhotic portal hypertension
* Acute on chronic liver failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in the incidence of first variceal bleed at 1 year. | 1 year

SECONDARY OUTCOMES:
Overall and bleed related Survival in all the 3 groups | 1 year
Bleed related Survival in all the 3 groups | 1 year
Improvement in Child-Turcotte-Pugh (CTP) score in all the 3 groups | 1 year
Improvement in Model for End Stage Liver Disease (MELD) score in all the 3 groups | 1 year
Incidence of Spontaneous Bacterial Peritonitis (SBP) in all the 3 groups | 1 year
Incidence of Acute Kidney Injury (AKI) in all the 3 groups | 1 year
Incidence of Shock in all the 3 groups | 1 year
Incidence of new ascites in all the 3 groups | 1 year
HVPG response at 1year in all the 3 groups | 1 year
Treatment related side effects in all the 3 groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tevethia HV, Pande A, Vijayaraghavan R, Kumar G, Sarin SK. Combination of carvedilol with variceal band ligation in prevention of first variceal bleed in Child-Turcotte-Pugh B and C cirrhosis with high-risk oesophageal varices: the 'CAVARLY TRIAL'. Gut. 2024 Oct 7;73(11):1844-1853. doi: 10.1136/gutjnl-2023-331181. PMID 39067870